CLINICAL TRIAL: NCT03923907
Title: Effectiveness of a Complex Exercise Intervention to Normalize Blood Pressure and Its Nocturnal Dipping in Patients With HyperTension in Primary Care: a Randomized-controlled Trial
Brief Title: Complex Exercise Intervention to Normalize Blood Pressure and Nocturnal Dipping in Patients With Hypertension
Acronym: END-HT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Lee Kam Pui, Clinical Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NTEC-2019-0264
Record Dates: First submitted 2019-04-16; First posted 2019-04-23 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Masking Description: The statistician will be masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EIM group (Experimental): patients with Hypertension (HT) will be recruited by a trained nurse when the patient attends the yearly to bi-yearly complication screening program called the risk assessment and management program (RAMP) program. This program is provided to all patients with HT, who are seen in the Government-funded primary care clinics in Hong Kong. The nurse will encourage the patient by motivational interviewing techniques and prescribe exercise. Combined exercise skills will be taught in the 12-week weekly exercise classes by certified physical trainers. Peer support is encouraged during and after the 12-week program. Regular feedback, prompting and problem solving will be provided by the nurse at 3m, 6m, and 12m. Exercise level will be monitored by validated wrist trackers to feedback participants, nurse and physical trainer by mobile apps and website. Resources to exercise will be made known to patients by apps, website and healthcare professionals.
  Interventions: Behavioral: EIM intervention group
- usual care (No Intervention): There is no extra intervention to patients allocated in this arm, except that they receive information and advice on lifestyle changes including benefits from exercise from the nurse at recruitment as stated above. Participants in both arms will have no changes in medication within the first 12-week to determine the BP difference between the two groups. In Hong Kong, patients have unlimited access to emergency department and general outpatient services. All patients with HT receive RAMP program counselling and screening every 1-2 years. These are not limited by the current trial.

INTERVENTIONS:
Behavioral: EIM intervention group — As in arm description
  Arms: EIM group

SUMMARY:
Background: Non-dipping hypertension(HT) (as defined by lack of decrease in systolic blood pressure (BP) by 10% during sleep) predicts cardiovascular events and mortality; however, there is a lack of evidence based treatment for non-dipping HT. While exercise is recommended to management HT, its effect on dipping status is not known. There is a lack of trials describing the relationship of exercise and blood pressure in Chinese.

Method: This will be a two-arm randomized controlled trial in which Chinese non-dippers (n= 198) will be randomized to an exercise program plus usual care or to usual care by stratified randomization. The randomization sequence is blinded to the investigators and allocation is disclosed only after valid consent. The exercise program utilizes various motivational techniques to enhance exercise maintenance.

ELIGIBILITY:
Inclusion Criteria:

* SBP non-dippers
* self-reported exercise intensity and duration less than the World Health Organization recommendation, which is exercise of moderate intensity less than 150minutes/week OR exercise of vigorous intensity of less than 75 minutes/week
* Used any mobile apps on their phone (because the intervention involve use of apps to monitor and remind regular exercise)

Exclusion Criteria

* Patients with diagnosed chronic obstructive lung disease and recent stroke (within last 12 months) because other evidence-proven and well-structured programmes are implemented for these patients in the hospital authority in Hong Kong
* Occupational drivers - because they need to hold their arm still during ABPM and this may be hazardous for drivers

  * night-time workers
  * diagnosed Obstructive Sleep Apnea
* Patients on anti-coagulants - because ABPM may induce bruises
* Patients on 3 or more medications for hypertension (on maximum tolerable doses) - these patients may have secondary HT and represent a different spectrum of organic diseases
* Patients with SBP >180mmHg or DBP >110mmHg - drug titration is not allowed during the 12-week program and these patients need early drug treatment
* Patient with DM - these patients will be arranged to have another EIM program especially designed for their DM.

  * Patients with active spinal cord compression or spinal radiculopathy because they may not be suitable to join some exercise
  * patients with atrial fibrillation are excluded because these patients have increased BP variability and may have different dipping behaviour
  * patients with metallic implants or pacemakers are excluded as they are not suitable for MRI
* To maximize safety of patients, patients who are relatively contraindicated according to AHA will also be excluded

  * acute myocardial infarction in last 6 months
  * ongoing angina
  * uncontrolled cardiac arrhythmia
  * acute diseases including known active endocarditis/acute pulmonary embolism, pulmonary infarction, deep vein thrombosis, acute aortic dissection, acute myocarditis
  * known aortic stenosis
  * known heart failure
  * known obstructive left main coronary artery stenosis
  * uncontrolled ventricular rates
  * complete heart block
  * known hypertrophic obstructive cardiomyopathy
  * mental impairment that limit co-operation
  * resting blood pressure with systolic blood pressure >180mmHg or diastolic blood pressure >110mmHg
  * known anemia with hemoglobin level less than 11gm/dL
  * known uncorrected electrolyte imbalance, and
  * known uncontrolled hyperthyroidism.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
systolic blood pressure(SBP) dipping status | at 12-week, after the EIM program
  as defined by a lack of SBP drop of more than 10% during sleep, as detected by ambulatory blood pressure measurements (ABPM)

SECONDARY OUTCOMES:
daytime, night-time, 24-h SBP, and DBP | baseline (before the 12-week program ), at 12 weeks and 12 months after recruitment
  as detected on ABPM discussed above
serum lipid profile | baseline (before the 12-week program ), at 12 weeks and 12 months after recruitment
  this includes serum total cholesterol, triglyceride , low-density lipoprotein and high-density lipoprotein
body mass index | baseline (before the 12-week program ), at 12 weeks, at 24 weeks and 12 months after recruitment
  weight and height will be combined to report BMI in kg/m^2
office blood pressure | baseline (before the 12-week program ), at 12 weeks, at 24 weeks and 12 months after recruitment
  office blood pressure will be measured 3 times and the last 2 will be averaged as the outcome
The Chinese version of international Physical Activity Questionnaire - short form (IPAQ-SF) | baseline (before the 12-week program ), at 12 weeks, at 24 weeks and 12 months after recruitment
  a validated questionnaire to detect exercise level; The questionnaire can provide the amount of time the participant spend on moderate or vigorous physical activities. The amount of energy spent can be calculated (metabolic equivalent of task; MET). For example, high level of exercise can be defined as a minimum total physical activity of at least 3000 MET minutes a week. The higher the MET, the higher the exercise level
systolic blood pressure(SBP) dipping status | measured at baseline and 12 months
  as defined by a lack of SBP drop of more than 10% during sleep, as detected by ambulatory blood pressure measurements (ABPM)
body fat percentage | baseline (before the 12-week program ), at 12 weeks, at 24 weeks and 12 months after recruitment
  body fat percentage
serum fasting glucose level | baseline (before the 12-week program ), at 12 weeks and 12 months after recruitment
  serum fasting glucose level
serum creatinine level | baseline (before the 12-week program ), at 12 weeks and 12 months after recruitment
  serum creatinine level that reflects renal function
waist circumference | baseline (before the 12-week program ), at 12 weeks and 12 months after recruitment
  waist circumference
serum high sensitive C-reactive protein | baseline (before the 12-week program ), at 12 weeks and 12 months after recruitment
  serum high sensitive C-reactive protein that reflect the degree of inflammation
MRI (proton density fat fraction) | baseline (before the 12 week program), at 12 weeks
  MRI liver to detect the degree of liver steatosis
Pittsburgh Sleep Quality Index(PSQI) | baseline (before the 12-week program ), at 12 weeks, at 24 weeks and 12 months after recruitment
  a validated questionnaire to detect sleep quality; possible "global" score include can range from 0 to 21. A global score of 5 or more indicates poor sleep quality; the higher the score, the worse the quality.
STOP-BANG (Snoring, Tiredness, Observed apnea, Blood pressure, Body mass index, Age, Neck circumference and Gender) questionnaire | baseline (before the 12-week program ), at 12 weeks, at 24 weeks and 12 months after recruitment
  a validated questionnaire to detect presence of sleep apnea; any 3 positive items from the 8 questions as having risk of OSA; the higher the number of positive items, the higher the risk

CONTACTS AND LOCATIONS:
Locations (1):
- Lek Yuen Clinic, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
Will be made available on request from investigators

REFERENCES:
- [Background] Lee EK, Zhang DD, Yip BH, Cheng J, Hui SS, Yu EYT, Leung M, Chu WCW, Mihailidou AS, Wong SY. Exercise Intervention to Normalize Blood Pressure and Nocturnal Dipping in HyperTensive Patients (END-HT): Protocol of a Randomized Controlled Trial. Am J Hypertens. 2021 Aug 9;34(7):753-759. doi: 10.1093/ajh/hpab019. PMID 33471104